CLINICAL TRIAL: NCT06402175
Title: Characteristics and Outcomes of Patients With Hematological Malignancies at Main Assuit University Hospital : A Single Centre Study
Brief Title: Characteristics and Outcomes of Patients With Hematological Malignancies
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Abdelslam Abudeif, Assistant Lecturer, Assiut University
Other Study IDs: Assiut Univesity
Record Dates: First submitted 2024-04-20; First posted 2024-05-07 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Haematologic Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: follow up — follow up

SUMMARY:
The pattern of hematological malignancies (HMs) in developing countries and developed countries differs. Among the different types of cancers, leukemia, lymphoma, and multiple myeloma appear to have greatly increased in frequency.

DETAILED DESCRIPTION:
The pattern of hematological malignancies (HMs) in developing countries and developed countries differs. Among the different types of cancers, leukemia, lymphoma, and multiple myeloma appear to have greatly increased in frequency. These malignancies are induced by genetic damage or mutation in somatic cells, which can result from environmental exposure to chemicals, ionizing radiation, and viral agents. Comparison of the incidence of HMs across geographic regions and time is complicated by the existence of different disease classification systems, and diagnostic criteria that vary by country, and even between hospitals and cancer registries (CRs) within a country.

Leukemia is a malignant neoplasm of hematopoietic stem cells characterized by diffuse replacement of bone marrow or peripheral blood by neoplastic cells; its etiology is obscure. Leukemia typing is based on how quickly the disease develops and progresses. Leukemia is either chronic or acute. Furthermore, leukemia typing is also based on the type of white blood cell that is affected. There are 4 common types of leukemia: acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), chronic myeloid leukemia (CML), and chronic lymphocytic leukemia (CLL). Most acute leukemias are classified as lymphoid or myeloid lineages via standard microscopic morphology, cytochemistry, and immunophenotyping. Previous studies have shown that there are important differences in the incidence of the various leukemia subtypes according to geography, race/ethnicity, age, and trend pattern, indicating that the subtypes may have different etiological factors and that comprehensive global assessment of leukemia patterns is warranted.

Lymphomas are a heterogenous group of diseases with differences in epidemiology, histology, and prognosis. The incidence of Hodgkin's lymphoma (HL) and nonHodgkin's lymphoma (NHL) is higher among males than females.

Multiple myeloma (MM) is included in the spectrum of diseases ranging from monoclonal gammopathy of unknown significance (MGUS) to plasma cell leukemia. Plasma cell proliferation usually results in extensive skeletal destruction, with osteolytic lesions, hypercalcemia, anemia, and occasionally plasma cell infiltration in different organs. Excessive production of a monoclonal (M) protein can lead to renal failure, hyperviscosity syndrome, or recurrent bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of Hematological malignancies (≥18 years)

Exclusion Criteria:

* patients who have started diagnosis and treatment for malignancy outside Assiut university.
* Age less than 18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: follow up of hematological malignancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
overall survival rate | 5 years
  Assessment of overall survival of hematological malignancies at Assiut university Hospital
  * Estimate rate of non-relapse mortality.
  * Estimate rate of complete remission.
  * Estimate rate of refractory disease.
  * Estimate the rate of relapsed diseases.

IPD SHARING:
Plan to Share IPD: No